

# **Evaluation of Post Operative Pain after obturation using two different types of sealers**

# (A Randomized Clinical Trial)

Research proposal submitted to Department of Endodontics, Faculty of Dentistry, British University in Egypt, in partial fulfillment of the requirements of master's degree in Endodontics

Submitted by

### Sara Tarek Mohamed Alsayed amin

Demonstrator in Endodontic Department Faculty of Dentistry, the British University in Egypt

(B.D.S. BUE, 2018)

#### Dr. Mohamed Medhat Kataia

Associate Professor of Endodontics

Acting Head of Department of Endodontics at the British University in Egypt

Faculty of Dentistry, British University in Egypt

## Dr. Hala Fayek Khalil

lecturer of Endodontics

Faculty of Dentistry, British University in Egypt

Department of Endodontics
Faculty of Dentistry
British University in Egypt
2021



## **Informed consent**

#### Research Title

Evaluation of the resulting pain after using different root canal adhesives in the root canals

#### Brief summary of the research:

Root canal treatment will be done for the patient and the root canals will be filled with different sealers – sealers based on calcium silicate or calcium phosphate or sealers based on resin, and then the resulting pain will be evaluated after treatment for the patient.

Principal Investigator: Dr. Sara Tarek Mohamed

Co-researchers: Prof. Mohamed Medhat Kataya and Dr. Hala Fayeq Khalil

Funding body: self-financing by researchers

#### General explanation of the situation and what will be done:

You suffer from severe decay in your teeth that led to inflammation of the roots, and you need root canal treatment to clean the canals and fill them with sealers . We are doing a study and we will use different types of sealers to evaluate the resulting pain afterwards.

#### Required of the participant in this study:

If you agree to participate with us in this study, you will be asked to attend one session at the university, and we will do the root canal treatment steps, and after the end of cleaning the root canals, and upon its completion, we will put a filling in the roots using different sealers and evaluate the resulting pain after filling 12 hours after treatment and 24 hours, 48 hours and 72 hours

Benefit: You will get free root canal treatment in the tooth you suffer from.

Treatment will be provided by specialized doctors.

The treatment will take place in the university's clinics with high capabilities, with sterile tools.

Get stuffing with new vital materials.

<u>Side effects:</u> Symptoms that may occur when doing root canal treatment, such as: failure of the procedure, which may require re-treatment, presence of a swelling, pain, inability to move the jaw for days, instrument separation inside the tooth, or a perforation (hole) in it that may lead to extraction of the tooth.

Possibility to accept or decline participation:

You are absolutely not obliged to participate, and you also have the right to withdraw from the study whenever you want after informing the responsible doctor without affecting your decision on the medical care you receive.

#### Who will know about your participation in the research:

The doctors responsible for the research, as well as the nurses assisting them, and you are free to inform whomever you want from your family and friends, and the information about your medical condition and treatment will be kept in a secure way, and it is not allowed to view it except for those responsible for the research.

If you have any other inquiries or if you want to ask any question during the study

You can direct it to Dr. Principal Investigator Dr. Sarah Tariq Muhammad, Tel: 01007434392

#### If you wish to raise any complaint during the study

Research number in the Ethics Committee:

You can direct it to Prof. Dr. Asmaa Yassin, Rapporteur of the Scientific Research Ethics Committee and Professor in the Department of Conservative Therapy at the British University, Tel: 01001912610

| I, the undersigned, acknowledge that I have read, understood and agree to participate in the stud |
|---|
| Participant's name: |
| phone number: |
| Participant address: |
| Study patient number: |
| Patient file number: National number: |
| History: |
| Witness Signature: Date: |
| Researcher's signature: Date: |